CLINICAL TRIAL: NCT04186663
Title: Pharmacokinetics of Advantage Arrest in Children
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Advantage Silver Dental Arrest, LLC (Industry)
Collaborators: University of California, San Francisco (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2019-06-23
Record Dates: First submitted 2019-11-28; First posted 2019-12-05 (Actual); Results first posted 2022-03-10 (Actual); Last update posted 2022-03-10 (Actual); Status verified 2021-05

CONDITIONS: Dental Caries
Keywords: child; pharmacokinetics; silver diamine fluoride
MeSH Terms: conditions — Dental Caries | interventions — silver diamine fluoride

STUDY DESIGN:
Intervention Model Description: Open label exposure--response study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Advantage Arrest (Experimental): 38% silver diamine fluoride, topical, 1 drop, single application
  Interventions: Drug: Silver Diamine Fluoride

INTERVENTIONS:
Drug: Silver Diamine Fluoride — 38% aqueous silver diamine fluoride [Ag(NH3)]2F, CAS RN 33040-28-7
  Other Names: Advantage Arrest

SUMMARY:
The purpose of this study is to characterize basic PK parameters (Cmax, t1/2, AUC) in healthy children to contribute to evidence for the safety of Advantage Arrest, consistent with Guidance for Industry--Exposure--Response Relationships (April 2003).

DETAILED DESCRIPTION:
This is a topical agent where the active ingredients are applied to the teeth and eventually swallowed and may be absorbed through the GI tract or excreted. Minimal amounts are absorbed through the oral mucosa. Serum concentrations of silver and fluoride will be be proportional to the dose of silver and fluoride administered topically to the teeth as part of Advantage Arrest. This is an open label exposure-response study with up to 50 healthy children ages 3-13 years of age. Subjects will be treated with Advantage Arrest and have one blood sample withdrawn at a randomly assigned time point. A minimum of 3 subjects per time point at 2,4,6,24,48,96 and 168 hours. Serum samples will be analyzed for F and Ag.

ELIGIBILITY:
Inclusion Criteria:

* Healthy.
* At least one carious lesion.

Exclusion Criteria:

* Oral mucositis
* Any ulcerative lesions
* Hypersensitivity to silver
* Hypersensitivity to fluoride.
* SDF treatment within 3 months.

Ages: 3 Years to 13 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 59 (Actual)
Dates: Start 2019-08-01 (Actual); Primary Completion 2020-03-31 (Actual); Study Completion 2020-03-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Hellene Ellenikiotis, DDS, Principal Investigator — University of California, San Francisco
Locations (1):
- University of California San Francisco Clinical and Translational Science Institute, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Advantage Arrest
Started | 59
Completed | 55
Not Completed | 4
Not completed — Lost to Follow-up | 1
Not completed — Unable to complete blood draw | 3

BASELINE CHARACTERISTICS:
Arm/Group | Advantage Arrest
Number analyzed (Participants) | 55
Age, Continuous [Mean (Standard Deviation); unit: years] | 7.7 (2.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 25
  Male | 30
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 24
  Not Hispanic or Latino | 25
  Unknown or Not Reported | 6
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 11
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 8
  White | 11
  More than one race | 0
  Unknown or Not Reported | 25
Region of Enrollment [Number; unit: participants]
  United States | 55
Weight (kg) [Mean (Standard Deviation); unit: kg] | 32.6 (16.5)

OUTCOME MEASURES:

1. Primary Outcome: Predicted Peak Serum Silver Concentration (Cmax)
Description: As only a single blood sample was obtained from each child, serum silver concentration versus time data were analyzed simultaneously using population pharmacokinetic analysis with nonlinear mixed effects modeling. The parameters estimated were the apparent volume of distribution (V/F) and apparent oral clearance (CL/F). The rate constant of absorption (ka) was fixed to 23.7 day-1. The predicted peak serum silver Cmax was calculated using Cmax = Dose/(V/F)*exp^(-k⋅tmax ), where k = (CL/F)/(V/F) and tmax = [ln(ka/k)]/(ka-k).
Time Frame: Based on data collected at 2, 4, 6, 24, 48, 96, and 168 hours post-SDF application
Population: Children who completed including blood draw
Measure: Mean (Standard Deviation); unit: ng/ml
Arm/Group | Advantage Arrest
Number analyzed (Participants) | 55
ng/ml | 17.8 (10.6)

2. Primary Outcome: Predicted Time to Peak Serum Silver Concentration (Tmax)
Description: As only a single blood sample was obtained from each child, serum silver concentration versus time data were analyzed simultaneously using population pharmacokinetic analysis with nonlinear mixed effects modeling. The parameters estimated were the apparent volume of distribution (V/F) and apparent oral clearance (CL/F). The rate constant of absorption (ka) was fixed to 23.7 day-1. The predicted time to peak concentration was calculated using tmax = [ln(ka/k)]/(ka-k), where k = (CL/F)/(V/F).
Time Frame: Based on data collected at 2, 4, 6, 24, 48, 96, and 168 hours post-SDF application
Population: Children who completed including blood draw
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Advantage Arrest
Number analyzed (Participants) | 55
hours | 5.1 (0.9)

3. Primary Outcome: Silver Half-life
Description: As only a single blood sample was obtained from each child, serum silver concentration versus time data were analyzed simultaneously using population pharmacokinetic analysis with nonlinear mixed effects modeling. The parameters estimated were the apparent volume of distribution (V/F) and apparent oral clearance (CL/F). The rate constant of absorption (ka) was fixed to 23.7 day-1. The half-life of silver was calculated using half-life = ln(2)/k, where k = (CL/F)/(V/F).
Time Frame: Based on data collected at 2, 4, 6, 24, 48, 96, and 168 hours post-SDF application
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Advantage Arrest
Number analyzed (Participants) | 55
days | 5.9 (4.7)

4. Secondary Outcome: Apparent Oral Clearance of Silver (CL/F)
Description: As only a single blood sample was obtained from each child, serum silver concentration versus time data were analyzed simultaneously using population pharmacokinetic analysis with nonlinear mixed effects modeling. The apparent oral clearance of silver (CL/F) was an estimated parameter.
Time Frame: Based on data collected at 2, 4, 6, 24, 48, 96, and 168 hours post-SDF application
Measure: Mean (Standard Deviation); unit: Liters/day
Arm/Group | Advantage Arrest
Number analyzed (Participants) | 55
Liters/day | 498 (496)

5. Secondary Outcome: Apparent Volume of Distribution of Silver (V/F)
Description: As only a single blood sample was obtained from each child, serum silver concentration versus time data were analyzed simultaneously using population pharmacokinetic analysis with nonlinear mixed effects modeling. The apparent volume of distribution (V/F) was an estimated parameter.
Time Frame: Based on data collected at 2, 4, 6, 24, 48, 96, and 168 hours post-SDF application
Measure: Mean (Standard Deviation); unit: Liters/day
Arm/Group | Advantage Arrest
Number analyzed (Participants) | 55
Liters/day | 2294 (1253)

6. Secondary Outcome: Serum Silver Exposure (AUC)
Description: Area under the curve of silver. As only a single blood sample was obtained from each child, serum silver concentration versus time data were analyzed simultaneously using population pharmacokinetic analysis with nonlinear mixed effects modeling. The parameters estimated were the apparent volume of distribution (V/F) and apparent oral clearance (CL/F). The rate constant of absorption (ka) was fixed to 23.7 day-1. The area under the curve was calculated using AUC = Dose/(CL/F).
Time Frame: Based on data collected at 2, 4, 6, 24, 48, 96, and 168 hours post-SDF application
Measure: Mean (Standard Deviation); unit: ng*day/mL
Arm/Group | Advantage Arrest
Number analyzed (Participants) | 55
ng*day/mL | 149 (140)

7. Other Pre Specified Outcome: Average Serum Fluoride Concentrations
Description: Overall average of measured serum fluoride concentrations at the various timepoints.
Time Frame: Collected at 2, 4, 6, 24, 48, 96, and 168 hours post-SDF application
Measure: Mean (Full Range); unit: ng/ml
Arm/Group | Advantage Arrest
Number analyzed (Participants) | 55
ng/ml | 15 [6 to 36]

ADVERSE EVENTS:
Time Frame: 168 h
Arm/Group | Advantage Arrest
All-Cause Mortality (participants affected / at risk) | 0/55
Serious Adverse Events (participants affected / at risk) | 0/55
Other Adverse Events (participants affected / at risk) | 0/55

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-06-23): https://cdn.clinicaltrials.gov/large-docs/63/NCT04186663/Prot_SAP_000.pdf